CLINICAL TRIAL: NCT05740423
Title: Anti-Seizure Medications Withdrawals After 2 Years of Seizure Remission
Brief Title: Standardization of Anti-Seizure Medications Withdrawals After Seizure Remission in Young Patients With Epilepsy
Acronym: ADORE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government); Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Min-Sun Yum, Professor, Asan Medical Center
Other Study IDs: HC20C0164; HC20C0164 (Other Grant/Funding Number: Korea Health Industry Development Institute)
Record Dates: First submitted 2023-01-03; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Epilepsy; Epilepsy in Children
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proper period of anti-seizure medication (ASM) treamtment is important for decreasing side effect of ASM and recurrence of seizure. We evaluate reliable risk factor analysis for safe withdrawal of ASM in children with epilepsy. Futhermore, we develop the scoring system for prediction of seizure recurrence to set the standard for safe withdrawal of ASM.

DETAILED DESCRIPTION:
The proper period of anti-seizure medication (ASM) treamtment is important for decreasing side effect of ASM and recurrence of seizure. We evaluate reliable risk factor analysis for safe withdrawal of ASM in children with epilepsy. Futhermore, we develop the scoring system for prediction of seizure recurrence to set the standard for safe withdrawal of ASM.

The enroll criteria as follow:

1. patients with epilepsy or acute provoked seizure accroding to the ILAE definition
2. patients who have been 2 years of seizure free with or without ASM

The patients with seizure recurrence during follow-up or end of follow-up period of 24 months will end this stutdy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Epilepsy or acute provoked seizure according to the ILAE guideline
* Patients with 2 years of seizure free periods

Exclusion Criteria:

* Uncertain diagnosis of epilepsy or acute provoked seizure
* Patients who do not want to participate in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Epilepsy or acute provoked seizure according to the ILAE guideline
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients umber of seizure recurrence | Up to 2 years
  Patients umber of seizure recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Min-Sun Yum, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea